CLINICAL TRIAL: NCT05327348
Title: The Efficacy of Perioperative Parenteral Ascorbic Acid in Reducing Oxidative Stress Among Patients Undergoing Free Flap Reconstructive Surgery: A Prospective Multicenter Randomized Controlled Pilot Trial
Brief Title: Effectiveness of IV Vitamin C in Reducing Oxidative Stress Associated With Free Flap Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MECID No,UMMC: 202086-8956; PV042-2021 (Other Grant/Funding Number: UMSC C.A.R.E); NMRR-21-1378-60482 (IIR) (Other: MOH Malaysia); USM/JEPeM/21070522 (Other: USM Malaysia)
Record Dates: First submitted 2022-03-28; First posted 2022-04-14 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Oxidative Stress; Ischemia-reperfusion Injury
Keywords: Free Flap Reconstructive Surgery; Perioperative Parenteral Ascorbic Acid
MeSH Terms: conditions — Reperfusion Injury | interventions — Ascorbic Acid; Saline Solution; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parenteral Ascorbic Acid (Experimental): Intravenous ascorbic acid 1 gram 8 hourly (3 grams per day) for 7 days
  Interventions: Drug: Intravenous Ascorbate
- 0.9% Normal Saline (Placebo Comparator): Intravenous 0.9% normal saline 10 mL 8 hourly for 7 days
  Interventions: Drug: Normal Saline 10 mL Injection

INTERVENTIONS:
Drug: Intravenous Ascorbate — Intravenous ascorbic acid 1 gram 8 hourly (3 grams per day) over 15 minutes for 7 days since pre-operative day 1 until post-operative day 5.
  Other Names: Ascorbic Acid Injection
  Arms: Parenteral Ascorbic Acid
Drug: Normal Saline 10 mL Injection — Intravenous 0.9% normal saline 8 hourly bolus infusion over 15 minutes for 7 days since pre-operative day 1 until post-operative day 5.
  Other Names: 0.9% Normal Saline
  Arms: 0.9% Normal Saline

SUMMARY:
Ischemia and reperfusion injury during free flap reconstructive surgery creates a state of increased oxidative stress that can adversely affect the flap outcomes. Ascorbic acid (AA) had been proven to have beneficial effect on end-organ protection and flap survival from ischemia-reperfusion injury via its antioxidant properties.

The investigators hypothesise that perioperative parenteral ascorbic acid treatment may reduce oxidative stress among participants undergoing free flap reconstructive surgery along with reduction in inflammatory markers, improved rate of flap viability and wound healing at both donor and recipient sites.

DETAILED DESCRIPTION:
Temporary cessation of blood supply to the flap tissues from clamping of donor vascular pedicle (ischemia) followed by restoration of flap tissue perfusion (reperfusion) after micro-anastomosis are inevitable in any free flap surgery. In combination, the ischemia and reperfusion process during free flap tissue transfers induce a state of increased oxidative stress, which may lead to complications such as flap failure and non-healing wounds at either donor or recipient sites. The negative impacts of which include additional wounds from flap loss, higher costs and increased duration of hospital stay.

Previous studies had demonstrated the beneficial effects of ascorbic acid in end-organ protection against ischemia and reperfusion injury. In addition, parenteral ascorbic acid has been shown to be remarkably safe even at high dose in both clinical and nonclinical models. Nonetheless, the data on efficacy of ascorbic acid in free flap survival in human is very limited.

The aims of this prospective, multicentre, double-blind, randomized, placebo-controlled pilot study are to measure the extent of oxidative stress in participants undergoing free flap reconstructive surgery before and after administration of parenteral ascorbic acid; and to evaluate its efficacy on modulation of inflammation, flap viability and wound healing.

Eligible participants will be randomized to receive 1 gram of parenteral ascorbic acid and 0.9% normal saline (as placebo) 8 hourly for 7 days (from pre-operative day 2 until post-operative day 5). Blood sampling will be performed on day 0 (pre-operative), day 3 (post-operative day 1) and day 5 (post-operative day 3) of intravenous ascorbic acid or placebo infusion for measurement of i) oxidative stress biomarkers, including isoprostane level, gene expression of glutamate-cystein ligase (GCL) and total glutathione level) ii) inflammatory markers, including leucocytes count and gene expression of TNF-α and IL-1. Post-operative outcomes of free flap surgery, up to post-operative 14 days, including flap viability, wound healing at both donor and recipient sites and duration of ICU and hospital stay will be evaluated.

The investigators estimate that a total sample of 28 participants (14 on each arm) will be necessary for 80% power to detect a 33% oxidative stress reduction with medium effect size (0.5) at 5% level of significance (α) between treatment (intravenous ascorbic acid) and placebo group (0.9% normal saline). A total of 34 participants are required to account for 20% of dropouts.

Primary analysis of this study utilizes an intention-to-treat approach and includes all randomized participants undergoing elective free flap reconstructive surgery. The mean difference between the baseline (pre-operative) and post-operative oxidative stress and inflammatory levels will be analyzed and compared between the intravenous ascorbic acid and placebo group using analysis of variance (ANOVA) for all normally distributed dataset whilst the non-parametric Kruskal-Wallis test is used, if otherwise. The effect size of such difference will be determined and compared. Subsequently, correlation between reduction of oxidative stress and post-operative flap outcomes in the intravenous ascorbic acid group will be evaluated. The secondary outcomes such as flap viability (percentage of flap necrosis), wound healing at both recipient and donor sites (percentage of wound dehiscence and percentage of skin graft failure to take/loss), duration of hospital and ICU stay and wound infection rate will be presented as mean with standard deviation (SD) or median with interquartile range (IQR) based on their normality distribution and are compared with Student's t-test or Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

- Adults (age 18 years and older, male or female) who are planned for elective free flap reconstructive surgery.

Exclusion Criteria:

* Hypersensitivity to vitamin C
* Oliguria (urine output <400mL/day) or anuria (urine output <100mL/day)
* Renal failure (serum creatinine level ≥175.0 %mol/L)
* Hemodialysis
* Renal calculi
* Thalassemia
* Glucose-6-phosphate dehydrogenase (G6PD) deﬁciency
* Unfit for surgery
* Pregnancy or lactating
* Hemochromatosis
* Hyperoxaluria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-09-25 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Oxidative stress biomarker: Plasma isoprostane level | Change from preoperative baseline level at day 5 of infusion (post-operative)
  Plasma isoprostane level will be analyzed using a competitive ELISA assay and expressed in unit of pg/ml.
Oxidative stress biomarker: Gene expression of glutamate-cystein ligase (GCL) | Change from preoperative baseline level at day 5 of infusion (post-operative)
  The expression of glutamate cysteine ligase (GCL) will be quantitated using real time quantitative polymerase chain reaction (qRT-CR). The differences in gene expression, expressed as fold-change, will be calculated using the 2 -DΔCt algorithm where GAPDH will be used as the housekeeping gene.
Oxidative stress biomarker: Total glutathione level | Change from preoperative baseline level at day 5 of infusion (post-operative)
  Total glutathione level (GSSG + GSH) will be determined using a Glutathione Assay Kit, which will be expressed in unit of µM.

SECONDARY OUTCOMES:
Inflammatory biomarkers levels: Leucocytes counts | Change from preoperative baseline level at day 5 of infusion (post-operative)
  Leucocytes count will be measured through flow cytometry White blood cells Differential Fluorescence (WDF) scattergram using Sysmex XN-10 (Sysmex Corporation TM , Kobe, Japan) and expressed in unit of X10^9/L.
Inflammatory biomarkers levels: Gene expression of TNF-α | Change from preoperative baseline level at day 5 of infusion (post-operative)
  The expression of TNF-α will be quantitated using real time quantitative polymerase chain reaction (qRT-CR). The differences in gene expression, expressed as fold-change, will be calculated using the 2 -DΔCt algorithm where GAPDH will be used as the housekeeping gene.
Inflammatory biomarkers levels: Gene expression of IL-1 | Change from preoperative baseline level at day 5 of infusion (post-operative)
  The expression of IL-1 will be quantitated using real time quantitative polymerase chain reaction (qRT-CR). The differences in gene expression, expressed as fold-change, will be calculated using the 2 -DΔCt algorithm where GAPDH will be used as the housekeeping gene.
Post-operative outcomes: Flap viability | From post-operative day 1 until day 14 (2 weeks)
  Flap viability is the survival of flap without tissue loss. For flap viability assessment, total flap loss is defined as complete necrosis (death) of flap (100% flap loss), whilst partial flap loss refers to incomplete necrosis of flap. By using simple tracing technique, the percentage of flap necrosis is calculated as:
  [Necrotic flap surface area (cm^2)/Total flap surface area (cm^2)] × 100%
Post-operative outcomes: Wound dehiscence | From post-operative day 1 until day 14 (2 weeks)
  Surgical wound dehiscence is defined as separation of the margins of a closed surgical incision that has been made in skin, with or without exposure or protrusion of underlying tissue, organs or implants. Wound dehiscence is assessed upon suture removal. It is categorized as either partial (1-99%) or complete (100%), depending on the depth/thickness of skin layers involvement. Partial wound dehiscence is defined as separation of wound edge up to level of epidermis and dermis layer of sutured wounds, whereas complete wound dehiscence refers to complete separation of wound edge involving the full thickness of skin. The percentage of wound dehiscence in relative to the total wound size is calculated.
Post-operative outcomes: Graft loss | From post-operative day 1 until day 14 (2 weeks)
  Skin graft recipient area is inspected at post-operative day 5 for assessment of graft take. Graft loss is categorized as partial (1-99%) or complete (100%). The percentage of skin graft failure to take/loss is calculated as:
  [Graft failure to take or loss surface area (cm^2)/Total skin graft area surface area (cm^2)] X 100%
Post-operative outcomes: Wound infection | From post-operative day 1 until day 14 (2 weeks)
  Wound infection is defined by presence of clinical sign and symptoms of infection associated with wound, including:
  i) Local signs: Erythema - localized or spreading (cellulitis); Pus/purulent or haemopurulent exudate; Abscess; Swelling/induration; Local warmth; Malodour; Crepitus; Dehiscence; Unexpected pain or tenderness.
  ii) Systemic signs: Malaise; Loss of appetite; Pyrexia or hypothermia; Tachycardia; Tachypnoea; Elevated C-reactive protein (CRP); Elevated or suppressed white blood cell count; Sepsis or Septic Shock.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Yii Shi Liang, MBBS, Principal Investigator — University of Malaya Medical Centre
Locations (3):
- Malaysia (3):
  - Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University of Malaya Medical Centre, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ballestin A, Casado JG, Abellan E, Vela FJ, Alvarez V, Uson A, Lopez E, Marinaro F, Blazquez R, Sanchez-Margallo FM. Ischemia-reperfusion injury in a rat microvascular skin free flap model: A histological, genetic, and blood flow study. PLoS One. 2018 Dec 27;13(12):e0209624. doi: 10.1371/journal.pone.0209624. eCollection 2018. PMID 30589864
- [Background] Schafer M, Werner S. Oxidative stress in normal and impaired wound repair. Pharmacol Res. 2008 Aug;58(2):165-71. doi: 10.1016/j.phrs.2008.06.004. Epub 2008 Jun 19. PMID 18617006
- [Background] Siemionow M, Arslan E. Ischemia/reperfusion injury: a review in relation to free tissue transfers. Microsurgery. 2004;24(6):468-75. doi: 10.1002/micr.20060. PMID 15378577
- [Background] Stepanovs J, Ozoliņa A, Rovīte V, Mamaja B, Vanags I. Factors Affecting the Risk of Free Flap Failure in Microvascular Surgery. Proc Latv Acad Sci Sect B Nat Exact, Appl Sci. 2016;70(6):356-364. doi:10.1515/prolas-2016-0039.
- [Background] Tsai MS, Huang CH, Tsai CY, Chen HW, Lee HC, Cheng HJ, Hsu CY, Wang TD, Chang WT, Chen WJ. Ascorbic acid mitigates the myocardial injury after cardiac arrest and electrical shock. Intensive Care Med. 2011 Dec;37(12):2033-40. doi: 10.1007/s00134-011-2362-6. Epub 2011 Sep 28. PMID 21953354
- [Background] Azari O, Kheirandish R, Azizi S, Farajli Abbasi M, Ghahramani Gareh Chaman S, Bidi M. Protective Effects of Hydrocortisone, Vitamin C and E Alone or in Combination against Renal Ischemia-Reperfusion Injury in Rat. Iran J Pathol. 2015 Fall;10(4):272-80. PMID 26351497
- [Background] Lee WY, Lee JS, Lee SM. Protective effects of combined ischemic preconditioning and ascorbic acid on mitochondrial injury in hepatic ischemia/reperfusion. J Surg Res. 2007 Sep;142(1):45-52. doi: 10.1016/j.jss.2006.08.043. Epub 2007 Jun 7. PMID 17559880
- [Background] Wang ZJ, Hu WK, Liu YY, Shi DM, Cheng WJ, Guo YH, Yang Q, Zhao YX, Zhou YJ. The effect of intravenous vitamin C infusion on periprocedural myocardial injury for patients undergoing elective percutaneous coronary intervention. Can J Cardiol. 2014 Jan;30(1):96-101. doi: 10.1016/j.cjca.2013.08.018. PMID 24365194
- [Background] Zaccaria A, Weinzweig N, Yoshitake M, Matsuda T, Cohen M. Vitamin C reduces ischemia-reperfusion injury in a rat epigastric island skin flap model. Ann Plast Surg. 1994 Dec;33(6):620-3. doi: 10.1097/00000637-199412000-00010. PMID 7880053
- [Background] Fowler AA 3rd, Syed AA, Knowlson S, Sculthorpe R, Farthing D, DeWilde C, Farthing CA, Larus TL, Martin E, Brophy DF, Gupta S; Medical Respiratory Intensive Care Unit Nursing; Fisher BJ, Natarajan R. Phase I safety trial of intravenous ascorbic acid in patients with severe sepsis. J Transl Med. 2014 Jan 31;12:32. doi: 10.1186/1479-5876-12-32. PMID 24484547
- [Background] Padayatty SJ, Sun AY, Chen Q, Espey MG, Drisko J, Levine M. Vitamin C: intravenous use by complementary and alternative medicine practitioners and adverse effects. PLoS One. 2010 Jul 7;5(7):e11414. doi: 10.1371/journal.pone.0011414. PMID 20628650
- [Background] Stephenson CM, Levin RD, Spector T, Lis CG. Phase I clinical trial to evaluate the safety, tolerability, and pharmacokinetics of high-dose intravenous ascorbic acid in patients with advanced cancer. Cancer Chemother Pharmacol. 2013 Jul;72(1):139-46. doi: 10.1007/s00280-013-2179-9. Epub 2013 May 14. PMID 23670640
- [Background] Hoffer LJ, Robitaille L, Zakarian R, Melnychuk D, Kavan P, Agulnik J, Cohen V, Small D, Miller WH Jr. High-dose intravenous vitamin C combined with cytotoxic chemotherapy in patients with advanced cancer: a phase I-II clinical trial. PLoS One. 2015 Apr 7;10(4):e0120228. doi: 10.1371/journal.pone.0120228. eCollection 2015. PMID 25848948